CLINICAL TRIAL: NCT06770426
Title: CompARing Between CO2 Phenylephrine and Phenylephrine Only Treatment in Patients With proGrEssing Cerebral infarctioN(CARBOGEN Trial)
Brief Title: CompARing Between CO2 Phenylephrine and Phenylephrine Only Treatment in Patients With proGrEssing Cerebral infarctioN
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2024-1415
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Acute Ischemic Stroke
Keywords: CO2; carbogen; phenylephrine; lacunar infarction; progressing stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke, Lacunar | interventions — carbogen; Phenylephrine

STUDY DESIGN:
Intervention Model Description: 1. The study is a single center, prospective, randomized, open-label trial with blinded end-point assessment (PROBE) design study.
  2. For the patients with progressing stroke, the carbogen + phenylphrine group and the phenylephrine only group will be randomized by 1: 1 through web-based app.
  3. Patients will be enrolled from February 2025 to September 2027 (based on the date of stroke).
  4. We will collect medical history, laboratory findings, neurological scores, and functional recovery.
  5. Functional recovery scores are performed by independent researchers in the blind state.
  6. All data is collected using e-CRF, and the image study will be anonymized and sent to the central adjudication.
  7. Central adjudication will review the image study.
Who Masked: Outcomes Assessor
Masking Description: Three months after discharge, the independence assessment will be perfomred by the researcher who don't know the patietns group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbogen + phenylephrine group (Experimental)
  Interventions: Drug: carbogen with or without phenyleprhine
- Phenylephrine group (Active Comparator)
  Interventions: Drug: phenylephrine

INTERVENTIONS:
Drug: carbogen with or without phenyleprhine — Patients will inhale carbogen gas for 10 minutes and rest for 50 minutes. All patients will recevive phenyleprhine to increase blood pressure. Start phenylephrine with 0.5 mg/hr and titrate upto 3.5 mg/hr or systolic blod pressure 200 mmHg.
  Arms: Carbogen + phenylephrine group
Drug: phenylephrine — All patients will recevive phenyleprhine to increase blood pressure. Start phenylephrine with 0.5 mg/hr and titrate upto 3.5 mg/hr or systolic blod pressure 200 mmHg.
  Arms: Phenylephrine group

SUMMARY:
Progressing stroke is associated poor functional outcome and neurological deficit.

Currently, no treatment for progressing stroke is recommended on the guideline.

Carbogen is a mixture of 5% CO2 with 95% O2. Carbogen is safe and it is used for the treatment of sudden sensory neural hearing loss or ocular ischemia.

CO2 dilate cerebral arteriole and concentration of CO2 is correlated with cerebral blood flow.

Increased cerebral blood flow following dilation of cerebral arteriole by CO2 might halt and revert progressing stroke.

Induced hypertension is alternative treatment of progressing stroke. Increasing blood pressure also induce cerebral blood flow. Phenylephrine is an α1 agonist, phenylephrine act on peripheral artery and little effect on cerebral artery or heart. Several studies reported that the effectiveness of phenylephrine on progressing stroke.

Therefore, this study will compare the effectiveness of carbogen + phenyleprhine versus phenlyephrine in progressing stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥20 years
* Anterior circulation progressing stroke
* Neurological worsening either 1 point in NIHSS score or MRC grade

Exclusion Criteria:

* Age under 20 years.
* Patients with cerebral infarction who are at risk of cerebral edema as determined by the investigator.
* Patients with Moyamoya disease.
* Patients with severe cerebrovascular reactivity (CVR) impairment due to cerebral vascular stenosis, making study participation challenging as determined by the investigator.
* Patients unable to undergo CO2 treatment (e.g., panic disorder, anxiety disorders, or other psychiatric conditions).
* Patients with hypersensitivity to phenylephrine.
* Patients with persistent bradycardia (heart rate < 50 bpm).
* Patients with a history of hemorrhagic stroke or at risk of cerebral hemorrhage.
* Patients with a pre-stroke modified Rankin Scale (mRS) score ≥ 2, indicating impaired functional independence.
* Patients ineligible for phenylephrine treatment due to any of the following:

Myocardial infarction or unstable angina within the past 3 months. Cardiac ejection fraction < 25%. Ventricular arrhythmia. Systolic blood pressure > 200 mmHg. Serum creatinine > 2 mg/dL. Pregnancy.

* Use of monoamine oxidase (MAO) inhibitors.
* Patients who do not consent to participate in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
percent improvement of NIHSS score in each group | 24 hours
  (baseline NIHSS score-post-treatment NIHSS score)/baseline NIHSS score×100
difference of NIHSS score in each group | 24 hours
  baseline NIHSS score-post-treatment NIHSS score
percent improvement of MRC score in each group | within 24 hours
  (baseline MRC score-post-treatment MRC score)/baseline MRC score×100
difference of MRC score in each group | difference of MRC score in each group
  baseline MRC score-post-treatment MRC score
Saftety outcome: Side effect | within 7 days
  Side effect (cerebral hemorrhage, myocardial infarction, Losing consciousness, difficulty breathing, dizziness, fatigue, headache, anxiety, etc)
Saftety outcome: discontinuing patients | within 7 days
  Number of discontinuing patients due to side effects

SECONDARY OUTCOMES:
Comparision between groups by percent improvement of NIHSS score | 24 hours
  (baseline NIHSS score-post-treatment NIHSS score)/baseline NIHSS score×100
Comparision between groups by differnece of NIHSS score | 24 hours
  baseline NIHSS score-post-treatment NIHSS score
Comparision between groups by percent improvement in MRC score | within 24 hours
  (baseline MRC score-post-treatment MRC score)/baseline MRC score×100
Comparision between groups by difference of MRC score | within 24 hours
  baseline MRC score-post-treatment MRC score
Functional independencec | 3 months after onset
  modifed Rankin score 0 to 2

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided